CLINICAL TRIAL: NCT07107425
Title: Accuracy of Non-Invasive Blood Pressure Monitoring During Laparoscopic Surgery in the Trendelenburg Position: A Prospective Error Grid Analysis
Brief Title: How Accurate Is Non-Invasive Blood Pressure Monitoring During Trendelenburg Laparoscopic Surgery?
Status: Not yet recruiting | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Kamil Darcin, Associate professor, Koç University
Other Study IDs: 2025.243.IRB2.109
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Non-Invasive Blood Pressure Monitoring in Trendelenburg Position
Keywords: Trendelenburg position; Laparoscopic surgery; Non-invasive blood pressure; Invasive arterial pressure; Error grid analysis; Hemodynamic monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Cohort: Adults (18 years and older) undergoing laparoscopic surgery in the Trendelenburg position who are already scheduled to receive invasive arterial blood pressure monitoring as part of routine clinical care. Participants will have paired invasive and non-invasive blood pressure measurements recorded during surgery for comparison using error grid analysis.

SUMMARY:
This study will test how accurate a blood pressure cuff is during certain types of surgery.

During some abdominal surgeries done with small tools and a camera (called laparoscopic surgery), doctors place patients in a head-down position called the Trendelenburg position. In this position, it may be harder for the blood pressure cuff on the arm to give correct readings. This study will compare the cuff's readings (non-invasive) with readings from a thin tube placed inside an artery (invasive), which is more accurate but also more risky and uncomfortable.

The researchers will use a method called error grid analysis to check how closely the cuff readings match the invasive ones. They hope to learn if the blood pressure cuff is accurate enough to be used safely in this kind of surgery. If it is, doctors may not need to use the invasive method as often.

People 18 years or older who are already going to have invasive blood pressure monitoring as part of their planned surgery can join the study. The study will collect blood pressure measurements about every 20 minutes during surgery, as well as basic information like age, weight, and what medicines are given.

DETAILED DESCRIPTION:
This is a prospective observational study designed to evaluate the clinical accuracy and reliability of non-invasive blood pressure (NIBP) monitoring in adult patients undergoing laparoscopic surgery in the Trendelenburg position. The accuracy of NIBP will be assessed by comparing it to invasive arterial blood pressure (IABP), which is considered the reference standard. The comparison will be performed using error grid analysis, a method that not only quantifies measurement differences but also categorizes the clinical risk of those discrepancies.

The Trendelenburg position, characterized by a head-down tilt of the patient, is frequently employed during gynecological and urological laparoscopic procedures to enhance surgical exposure. However, this positioning alters hemodynamic physiology and may influence peripheral blood pressure measurements. Previous evaluations of NIBP in this context have primarily relied on Bland-Altman analysis, which measures statistical agreement but does not assess the potential clinical consequences of disagreement between methods.

Error grid analysis overcomes this limitation by mapping paired NIBP and IABP values into predefined risk zones (A-E), based on their potential to affect clinical decision-making. Zone A reflects acceptable agreement with no risk of incorrect treatment, whereas Zones B through E indicate increasing levels of clinical risk.

In this study, NIBP and IABP will be measured simultaneously every 20 minutes throughout the procedure. The proportion of measurements falling within each error grid zone will be calculated. If fewer than 90% of the paired measurements fall within Zone A, NIBP will be considered insufficiently reliable for use in this surgical context without concurrent invasive monitoring.

A pilot study of five patients was conducted to estimate the intracluster correlation coefficient and design effect, which informed the final sample size calculation. Based on these preliminary data, a total of 100 patients is estimated to provide adequate statistical power to evaluate the primary outcome with 95% confidence and a 5% margin of error.

The study will also document intraoperative variables that may affect blood pressure measurement accuracy, including the use of vasoactive infusions. These data may provide insight into subgroups where NIBP reliability is particularly limited or acceptable.

The findings of this study may inform future monitoring protocols and could reduce unnecessary use of invasive lines in appropriately selected patients, improving patient safety and comfort while maintaining clinical accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled to undergo laparoscopic surgery in the Trendelenburg position
* Will receive invasive arterial blood pressure monitoring as part of routine clinical care

Exclusion Criteria:

* Has peripheral artery disease
* Has congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from adult patients scheduled for laparoscopic surgery in the Trendelenburg position at Koç University Hospital, a tertiary care academic medical center in Istanbul, Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of Paired Systolic Blood Pressure Measurements Within Zone A of the Error Grid | Intraoperative period (measurements taken every 20 minutes during surgery)
  The percentage of systolic non-invasive blood pressure (NIBP) measurements that fall within Zone A of the consensus error grid with calibrated risk zones, as described by Saugel et al.[1]. Zone A represents measurement pairs with no risk of leading to inappropriate clinical decisions, based on comparison with simultaneously recorded systolic invasive arterial blood pressure values. Systolic NIBP measurements will be considered acuurate if 90% or more of the paired values fall within Zone A.
  1. Saugel B, Grothe O, Nicklas JY. Error Grid Analysis for Arterial Pressure Method Comparison Studies. Anesth Analg. 2018 Apr;126(4):1177-1185
Proportion of Paired Mean Arterial Pressure (MAP) Measurements Within Zone A of the Error Grid | Intraoperative period (measurements taken every 20 minutes during surgery)
  The percentage of non-invasive mean arterial pressure (MAP) measurements that fall within Zone A of the consensus error grid with calibrated risk zones, as described by Saugel et al.[1]. Zone A represents measurement pairs with no risk of leading to inappropriate clinical decisions, based on comparison with simultaneously recorded invasive MAP values. Non-invasive MAP measurements will be considered accurate if 90% or more of the paired values fall within Zone A.
  1. Saugel B, Grothe O, Nicklas JY. Error Grid Analysis for Arterial Pressure Method Comparison Studies. Anesth Analg. 2018 Apr;126(4):1177-1185

SECONDARY OUTCOMES:
Distribution of Paired Systolic Blood Pressure Measurements Across All Error Grid Zones (A-E) | Intraoperative period (measurements taken every 20 minutes during surgery)
  The percentage of paired systolic blood pressure measurements that fall into each zone (A, B, C, D, E) of the consensus error grid. Error grid zones reflect the clinical risk of acting on the non-invasive measurement:
  Zone A: No risk Zone B: Low risk Zone C: Moderate risk Zone D: Significant risk of undertreatment Zone E: Significant risk of overtreatment The distribution will be reported as the percentage of all paired measurements falling into each zone.
Distribution of Paired Mean Arterial Pressure (MAP) Measurements Across All Error Grid Zones (A-E) | Intraoperative period (measurements taken every 20 minutes during surgery)
  the percentage of paired mean arterial pressure (MAP) measurements that fall into each zone (A through E) of the consensus error grid. Error grid zones reflect the clinical risk of acting on the non-invasive measurement: Zone A: No risk Zone B: Low risk Zone C: Moderate risk Zone D: Significant risk of undertreatment Zone E: Significant risk of overtreatment The distribution will be reported as the percentage of all paired measurements falling into each zone.
Effect of Antihypertensive Medication Use on the Accuracy of Systolic NIBP Measurements | Intraoperative period (measurements taken every 20 minutes during surgery)
  This outcome compares the likelihood that individual systolic non-invasive blood pressure (NIBP) measurements fall within Zone A of the consensus error grid between participants who use antihypertensive medications and those who do not. Zone A indicates values that would not lead to inappropriate clinical decisions.
  To account for the fact that multiple blood pressure measurements are collected from each participant, the analysis will use mixed-effects logistic regression. This model includes a random effect for each participant to account for the correlation among repeated measurements within the same individual.
Effect of Antihypertensive Medication Use on the Accuracy of Mean Arterial Pressure (MAP) NIBP Measurements | Intraoperative period (measurements taken every 20 minutes during surgery)
  This outcome compares the likelihood that individual non-invasive mean arterial pressure (MAP) measurements fall within Zone A of the consensus error grid between participants with and without antihypertensive medication use. Zone A represents measurement pairs that are clinically acceptable.
  To account for the fact that multiple blood pressure measurements are collected from each participant, the analysis will use mixed-effects logistic regression. This model includes a random effect for each participant to account for the correlation among repeated measurements within the same individual.

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Darcin, MD, Study Director — Koç University School of Medicine
Locations (1):
- Koc University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) that underlie the results of the study will be shared. These data will be made publicly available through the Zenodo repository following study completion and publication.
Supporting Information: Study Protocol
Time Frame: Beginning at the time of the first publication of study results, with no end date.
Access Criteria: The anonymized individual participant data (IPD) and supporting documentation will be openly available to the public via the Zenodo data repository. No proposal, request, or data use agreement is required. Researchers may download the dataset directly from Zenodo upon publication. The data are intended for secondary analysis, validation of findings, or meta-research. A citation to the original study publication and dataset DOI is requested when using the data.
URL: https://zenodo.org/

REFERENCES:
- [Background] Saugel B, Grothe O, Nicklas JY. Error Grid Analysis for Arterial Pressure Method Comparison Studies. Anesth Analg. 2018 Apr;126(4):1177-1185. doi: 10.1213/ANE.0000000000002585. PMID 29239945